CLINICAL TRIAL: NCT07358975
Title: Prediction of Complications in Patients Undergoing Surgical Treatment of Hepatic Tumors
Brief Title: Prediction of Complications in Hepatic Tumors
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Danish Cancer Society (Other)
Responsible Party: Principal Investigator, Hans-Christian Pommergaard, Associate professor, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GSA-HEPSURU-RH
Record Dates: First submitted 2025-12-05; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-11

CONDITIONS: Hepatic Tumors
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: The aim of this study is to evaluate the diagnostic accuracy of [99mTc] Tc-GSA SPECT/CT in quantifying liver function in European patients with hepatic tumors. For accomplish this objective, in 2022, the Department of Clinical Physiology and Nuclear Medicine at Rigshospitalet optimized the in-house production of [99mTc] Tc-GSA under European regulations, and in April 2025, received approval from the Danish Medicines Agency for its clinical use. The compassionate permit allows the use of [99mTc] Tc-GSA for preoperative evaluation of regional liver function in the part of the liver that is preserved after liver resection due to malignant liver disease (primary liver cancer, primary biliary cancer and colorectal liver metastases). This study will explore the benefits of using [99mTc] Tc-GSA in combination with SPECT/CT in patients with a confirmed or suspected diagnosis of hepatic tumor (benign ot malignant) and a planned local treatment (resection and/or ablation).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All participants (Experimental)
  Interventions: Diagnostic Test: [99mTc] Tc-GSA SPECT/CT

INTERVENTIONS:
Diagnostic Test: [99mTc] Tc-GSA SPECT/CT — To evaluate preoperative liver function using [99mTc] Tc-GSA SPECT/CT, participants will receive an intravenous injection of 185 MBq/3 mg [99mTc] Tc-GSA through a peripheral vein. SPECT imaging will be performed 20 minutes after tracer injection.

SUMMARY:
Liver failure is one of the most severe complications in patients undergoing liver surgery for hepatic malignancies. However, it can be predicted through preoperative assessment of liver function. Technetium-99m galactosyl human serum albumin ([99mTc] Tc-GSA), combined with single-photon emission computed tomography fused with computed tomography ([99mTc] Tc-GSA SPECT/CT), is widely used in Asia due to its superiority in predicting postoperative liver failure. Unfortunately, its clinical use in Western countries remains limited due to concerns about disease transmission.

In 2022, the Department of Clinical Physiology and Nuclear Medicine at Rigshospitalet optimized the in-house production of [99mTc] Tc-GSA under European regulations, and in April 2025, received approval from the Danish Medicines Agency for its clinical use. This study aims to evaluate, for the first time, the diagnostic accuracy of [99mTc] Tc-GSA SPECT/CT in quantifying liver function in European patients with hepatic tumors.

Hypothesis: [99mTc] Tc-GSA SPECT/CT is capable of and superior to indocyanine green clearance test (ICG), Child-Pug score, Model for End-Stage Liver Disease (MELD) score, and ultrasound elastography in quantifying liver function and predicting surgical outcomes in a Danish cohort of patients with liver tumors. Perceived quality of life may be associated with postoperative complications. However, postoperative complications and survival can be more accurately predicted when quality of life is assessed in combination with preoperative liver function and clinical conditions.

Objectives

Primary objectives:

1. To evaluate the correlation between [99mTc] Tc-GSA SPECT/CT and established liver function assessments, including ICG clearance, Child-Pugh score, MELD score, and ultrasound elastography.
2. To compare the discriminative ability of [99mTc] Tc-GSA SPECT/CT with existing liver function tests in predicting postoperative complications.

   Secondary objectives:
3. To assess the correlation of [99mTc] Tc-GSA SPECT/CT, ICG clearance, Child-Pugh score, MELD score, and ultrasound elastography with postoperative outcomes.
4. To develop and internally validate a multivariable predictive model combining the best predictive liver function test with preoperative clinical characteristics to predict postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

Adults over 18 years who have the capacity to act, with a confirmed or suspected diagnosis of one or more hepatic tumors and a planned local treatment proposed by a multidisciplinary team of specialists, specifically those:

1. Patients undergoing major liver resection (FLR < 40%).
2. Patients undergoing minor resections or open/laparoscopic ablations with a risk of impaired liver function, defined by at least one of the following:

   * Histological diagnosis of liver cirrhosis or fibrosis (Meta-analysis of Histological Data in Viral Hepatitis scoring system [METAVIR] score 1 to 4).
   * Radiological signs of cirrhosis.
   * Preoperative chemotherapy.
   * Known liver disease associated with cirrhosis: metabolic dysfunction-associated steatohepatitis, chronic infection with hepatitis B or C, primary sclerosing cholangitis, primary biliary cholangitis, and autoimmune hepatitis.

Exclusion Criteria:

* History of hypersensitivity to Technetium-99m or albumin
* Diagnosis of pulmonary hypertension,
* Pregnant or breastfeeding individuals. For fertile women, non-pregnancy must be confirmed by a negative pregnancy test. No contraception methods are required after the study due to the short radioactive half-life of the IMP.
* Patients under 18 years old or unable to make autonomous care decisions.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Correlation between [99mTc] Tc-GSA SPECT/CT parameters and ICG clearance | Once before receiving the planned treatment for a hepatic tumor.
  The correlation between quantitative liver uptake parameters derived from [99mTc] Tc-GSA SPECT/CT and indocyanine green (ICG) clearance will be assessed using Pearson's/Spearman's rank correlation coefficient.
  [99mTc] Tc-GSA SPECT/CT units: Liver function test expresed in Uptake Index (UI) and percentage of total liver volume (FLR%).
  Indocyanine green (ICG) clearance units: Liver function test reported as: 1.- ICG retention ratio after 15 min (ICGR15), unit: percentage (%) 2.- Rate constant (k) of ICG indicator-dilution curve (KICG), unit: min-1 3.- Plasma dis-appearance rate of ICG (PDRICG), unit: % min-1.
Correlation between [99mTc] Tc-GSA SPECT/CT parameters and Child-Pugh score | Once before receiving the planned treatment for a hepatic tumor.
  The correlation between quantitative [99mTc] Tc-GSA SPECT/CT-derived liver function parameters and Child-Pugh score will be assessed using Pearson's/Spearman's rank correlation coefficient.
  [99mTc] Tc-GSA SPECT/CT units: Uptake Index (UI) and percentage of total liver volume (FLR%).
  Child-Pug score description and units: : Scoring system that estimates cirrhosis severity. It classifies patients into three categories: A - good hepatic function, B - moderately impaired hepatic function, and C - advanced hepatic dysfunction.
Correlation between [99mTc] Tc-GSA SPECT/CT parameters and the Model for End-Stage Liver Disease (MELD) score | Once before receiving the planned treatment for a hepatic tumor.
  he correlation between quantitative [99mTc] Tc-GSA SPECT/CT-derived liver function parameters and MELD score will be assessed using Pearson's/Spearman's rank correlation coefficient.
  [99mTc] Tc-GSA SPECT/CT units: Uptake Index (UI) and percentage of total liver volume (FLR%).
  MELD score definition and units: The Model for End-Stage Liver Disease (MELD) is a prognostic score to measure the severity of liver failure. The MELD score is based on results from five blood tests: Bilirubin, Creatinine, Internal normalized ratio (INR), Serum sodium, and Albumin. The MELD score ranges from 6 to 40, and quantifies end-stage liver disease for transplant planning. The higher the score, the more severe the disease.
Correlation between [99mTc] Tc-GSA SPECT/CT parameters and liver stiffness measured by ultrasound elastography | Once before receiving the planned treatment for a hepatic tumor.
  The correlation between quantitative [99mTc] Tc-GSA SPECT/CT-derived liver function parameters and liver stiffness measured by ultrasound elastography will be assessed using Pearson's/Spearman's rank correlation coefficient.
  99mTc] Tc-GSA SPECT/CT units: Uptake Index (UI) and percentage of total liver volume (FLR%) Ultrasound elastography: kilopascals (kPa)
Discriminative ability of [99mTc] Tc-GSA SPECT/CT compared with standard liver function tests to predict major postoperative complications | Once after the completion of 90-day follow-up.
  The discriminative ability of [99mTc]Tc-GSA SPECT/CT to predict major postoperative complications (Clavien-Dindo grade ≥ III) will be compared with standard liver function tests, including ICG clearance, Child-Pugh score, MELD score, and ultrasound elastography (units and definitions have been previously described).
  The Clavien-Dindo classification ranks the severity of surgical complications and consists of seven grades (I, II, IIIa, IIIb, IVa, IVb, and V). Complications of grade ≥ III will be considered major.
  Discriminative performance will be assessed using the area under the receiver operating characteristic curve (AUC) for each test. AUCs will be compared using DeLong's test.

SECONDARY OUTCOMES:
Association of [99mTc] Tc-GSA, ICG, Child-Pugh, MELD, and ultrasound elastography with 90-day mortality | Once during the final analysis after completion of 90-day follow-up.
  A regression model will be run between the variables. Parameters derived from [99mTc] Tc-GSA, ICG, Child-Pugh, MELD, and ultrasound elastography will be treated as independent variables, while 90-day mortality will be treated as binary and dependent variable.
  Units for [99mTc] Tc-GSA, ICG, Child-Pugh, MELD, and ultrasound elastography has been described before.
  90-day mortality categories: yes, no.
Association of [99mTc] Tc-GSA, ICG, Child-Pugh, MELD, and ultrasound elastography with post-hepatectomy liver failure | Once during the final analysis after completion of 90-day follow-up.
  A regression model will be run between the variables. Parameters derived from [99mTc] Tc-GSA, ICG, Child-Pugh, MELD, and ultrasound elastography will be treated as independent variables, while post-hepatectomy liver failure will be treated as binary and dependent variable.
  Units for [99mTc] Tc-GSA, ICG, Child-Pugh, MELD, and ultrasound elastography has been described before.
  Post-hepatectomy liver failure categories: yes, no
Association of [99mTc] Tc-GSA, ICG, Child-Pugh, MELD, and ultrasound elastography with length of stay. | Once during the final analysis after completion of 90-day follow-up.
  A regression model will be run between the variables. Parameters derived from [99mTc] Tc-GSA, ICG, Child-Pugh, MELD, and ultrasound elastography will be treated as independent variables, while length of stay. will be treated as dependent variable.
  Units for [99mTc] Tc-GSA, ICG, Child-Pugh, MELD, and ultrasound elastography has been described before.
  Units for length of stay: days
Association of [99mTc] Tc-GSA, ICG, Child-Pugh, MELD, and ultrasound elastography with readmission. | Once during the final analysis after completion of 90-day follow-up.
  A regression model will be run between the variables. Parameters derived from [99mTc] Tc-GSA, ICG, Child-Pugh, MELD, and ultrasound elastography will be treated as independent variables, while readmision will be treated as binary and dependent variable.
  Units for [99mTc] Tc-GSA, ICG, Child-Pugh, MELD, and ultrasound elastography has been described before.
  Readmision: yes, no
Model development and internal validation of a multivariable predictive model combining the most accurate liver function test with preoperative clinical factors (frailty, sarcopenia, grip strength, age, sex, etc.) to predict complications. | Once during the final analysis after completion of 90-day follow-up.
  The model performance will be assessed using penalized regression with discrimination, calibration, and bootstrap validation.

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No